CLINICAL TRIAL: NCT02430506
Title: A Phase I Randomized Placebo-controlled Double-blind Study to Evaluate Safety and Immunogenicity of AERAS-402 Administered in HIV-negative, BCG-vaccinated, QuantiFERON®-TB Gold (+) and QuantiFERON®-TB Gold (-) Adults Without Evidence of Tuberculosis.
Brief Title: A Study to Evaluate Safety and Immunogenicity of AERAS-402 Administered in HIV-negative, BCG-vaccinated, QFT (+) and (-) Adults Without Evidence of TB
Acronym: C-012-402
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aeras (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C-012-402
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — AERAS-402

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 1.0 mL sterile buffer administered by intramuscular (IM) injection to deltoid area on days 0 and 56.
  Interventions: Biological: Placebo
- AERAS-402 (Experimental): 1.0 mL containing 3 x 10^10 vp/mL suspended in 20 mM Tris buffer, 2 mM MgCl2, 25 mM NaCl, 10% w/v sucrose, 0.02% w/v PS-80 (polysorbate-80, non-animal source) and water. Administered intramuscular (IM) injection to deltoid area on days 0 and 56.
  Interventions: Biological: AERAS-402

INTERVENTIONS:
Biological: Placebo — This is the identical buffer solution in which AERAS-402 is formulated.
  Arms: Placebo
Biological: AERAS-402 — Given to 8 participants that were QFT-G(-) at screening and 8 participants that were GFT-G(+) at screening.
  Arms: AERAS-402

SUMMARY:
The available live tuberculosis vaccine Bacillus Calmette-Guérin (BCG) provides incomplete protection against pulmonary tuberculosis. For unknown reasons, a BCG revaccination or "booster", while not toxic, does not provide much additional protection. AERAS-402 presents tuberculosis antigens in the setting of a new, live, replication deficient adenovirus vaccine that may increase T cell immunity and thus protection from tuberculosis. Since BCG-vaccinated individuals are the population for which AERAS-402 might be indicated, AERAS-402 will be administered to individuals in Kenya who have already been vaccinated with BCG.

DETAILED DESCRIPTION:
This Phase I study will be conducted as a double-blind, randomized, placebo-controlled study in 20 healthy adult subjects. The study will enroll 10 subjects who are QFT-G positive at screening and 10 subjects who are QFT-G negative at screening. Within QFT-G group, subjects will be randomized to receive AERAS-402 or placebo in a ratio of 4:1. One dose level of AERAS-402 (3 x 10^10 vp) will be investigated in this study. All subjects will receive a single dose of study vaccine (AERAS-402 or placebo) on Study Day 0 and a second dose of study vaccine (AERAS-402 or placebo) on Study Day 56. All vaccinations will be administered by IM injection into the deltoid muscle.

The sample size was selected as adequate for preliminary safety evaluations and initial immunogenicity reviews for this phase study, rather than for statistical reasons. If no serious adverse events are observed in 16 subjects who receive AERAS-402, the upper bound of the 95% confidence interval on the rate of serious adverse event occurrence is 17.1 percent.

The selection of AERAS-402 dose level for evaluation in this study was derived from animal studies and based on the safety profile for the completed and ongoing clinical studies in the U.S. and South Africa.The total duration of follow-up is 182 days for each subject with a total of eleven follow-up clinic visits. The study is planned at a single site in Kisumu, Kenya.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female
2. Is age 18 through 45 years on Study Day 0
3. Has completed the written informed consent process
4. Had BCG vaccination at least 5 years ago, documented through medical history or presence of scar
5. Females: Ability to avoid pregnancy from 28 days prior to administration of the study vaccine through the end of the study.
6. Has general good health, confirmed by medical history and physical examination.
7. Has Body Mass Index (BMI) between 18 and 30 (wt./ht.2) by nomogram
8. Has ability to complete follow-up period of 182 days as required by the protocol
9. Is able and willing to commit to avoiding elective surgery for the duration of the study.
10. Is able and willing to stay in contact with the study site for the duration of the study.
11. Has completed simultaneous enrollment in Aeras Vaccine Development Registry Protocol.

Exclusion Criteria:

1. Acute illness on the day of randomization.
2. Fever ≥37.5°C on the day of randomization.
3. Evidence of any significant active infection on the day of randomization.
4. Used immunosuppressive medication within 45 days before entry into the study (inhaled and topical corticosteroids are permitted).
5. Received immunoglobulin or blood products within 45 days before entry into the study.
6. Received any investigational drug therapy or vaccine within 182 days before the first dose of study vaccine in this protocol.
7. Received any standard vaccine within 45 days before the first dose of study vaccine in this protocol, through the last study visit (the use of licensed drugs or vaccines medically indicated during the study is permitted).
8. Received any adenovector based vaccine previously.
9. Current chronic drug therapy including hormones such as thyroxin, insulin, etc. (Estrogen and progesterone replacement and contraceptives are permitted)
10. History or laboratory evidence of any past, present or future possible immunodeficiency state which will include, but is not limited to, any laboratory indication of HIV-1 infection.
11. History of allergic disease or reactions likely to be exacerbated by any component of the study vaccine.
12. Previous medical history that may compromise the safety of the subject in the study.
13. Evidence of a new acute illness that may compromise the safety of the subject in the study.
14. Pregnant or lactating/nursing females.
15. Evidence of chronic hepatitis including a positive test for hepatitis B core antibody, or hepatitis C antibody.
16. Inability to discontinue daily medications except contraceptives during the study.
17. History of alcohol or drug abuse within the past 2 years.
18. Tobacco or cannabis smoking three or more days per week
19. Positive urine test for illicit drugs (opiates, cocaine, amphetamines).
20. History or evidence of any systemic disease on physical examination or any acute or chronic illness that may interfere with the evaluation of the safety or immunogenicity of the vaccine, including axillary lymphadenopathy
21. History or evidence (including chest X-ray) of active or past tuberculosis
22. Abnormal hemoglobin, hematocrit, white blood cell count, absolute neutrophil count, absolute lymphocyte count, PT, PTT, GGT, ALT, AST, total bilirubin, ALP, and creatinine drawn within 36 hours of randomization. CPK must be drawn but the CPK value is not an exclusion criteria.
23. History of high risk sexual behaviors.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety of AERAS-402 in healthy, HIV-negative, BCG-vaccinated, QuantiFERON®-TB Gold In-Tube test (QFT-G)(+) and QFT-G(-) adults without evidence of tuberculosis disease in Kenya. | Day 0 thru Day 182
  Collection of solicited and unsolicited adverse events.

SECONDARY OUTCOMES:
Immunogenicity profile of AERAS-402 in healthy, HIV-negative, BCG-vaccinated, QFT-G(+) and QFT-G(-) adults without evidence of tuberculosis disease in Kenya. | Day 0 thru day 182
  Percentage of CD4 and CD8 T cells that produce any of three cytokines (IFN-γ, TNF-α, and/or IL-2) or a combination of the three cytokines simultaneously.

CONTACTS AND LOCATIONS:
Overall Officials: Doug Walsh, MD, Principal Investigator — U. S. Army Medical Research Unit- Kenya
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya

REFERENCES:
- [Background] Walsh DS, Owira V, Polhemus M, Otieno L, Andagalu B, Ogutu B, Waitumbi J, Hawkridge A, Shepherd B, Pau MG, Sadoff J, Douoguih M, McClain JB; Aeras C-012-402 Study Team. Adenovirus type 35-vectored tuberculosis vaccine has an acceptable safety and tolerability profile in healthy, BCG-vaccinated, QuantiFERON((R))-TB Gold (+) Kenyan adults without evidence of tuberculosis. Vaccine. 2016 May 5;34(21):2430-2436. doi: 10.1016/j.vaccine.2016.03.069. Epub 2016 Mar 26. PMID 27026148